CLINICAL TRIAL: NCT03292068
Title: Children Recovering From Tonsil Surgery Following Day Surgery
Brief Title: Children Recovering From Tonsil Surgery
Acronym: TONIST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Helena Rosén, PhD, Principal investigator, Lund University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TONIST
Record Dates: First submitted 2017-06-15; First posted 2017-09-25 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Tonsillitis
MeSH Terms: conditions — Tonsillitis | interventions — Acupuncture Therapy; Acupressure; Egg Yolk

STUDY DESIGN:
Intervention Model Description: Triangulation design will be used including both qualitative and quantitative methods. All the intervention groups will receive usual care in combination with a special intervention. The control group will only receive usual care. In the study the three interventions will be performed at one hospital each.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupuncture, acupressure (Experimental): Intervention with Pyonex-needles & Usual care; applied to the acupoints LI4 , LI11, PC6 and ST36 bilaterally before surgery. Pyonex needles are embedded in a 2 mm round plastic piece sitting on a round, skin friendly patch of about 8 mm in diameter. The patch can remain for seven days. The needle can be stimulated by gently touches the plastic bubble by the patch.
  Intervention Acupressure & Usual care; a 'kulplåster (1.5 mm a ball on a small piece of adhesive tape) both ears before postoperative drug administration. Kulplåster can remain for ten days or until they fall off. Children and their parents will be asked to fill in a diary of when the needle is stimulated, for what reason and when the symptoms are alleviated. In the diary is also filled in on the kulplåster remains.
  Interventions: Combination Product: Acupuncture, acupressure
- Timbal diet (Experimental): Timbal diet including ice cream & Usual care.The specially designed diet, originally made for patients suffering of dysphagia, named "timbalkost" will be used. The specially designed food/diet, "timbalkost" will be given as lunch and dinner. The consistency of timbalkost is smooth. It does not require more thorough processing of the mouth. As a snack, a protein-enriched ice cream, made with egg yolks and cream, will be made available. The food will be given to the child for 3-7 days depending on how quickly the child can return to normal food. A powder that jellify liquids to facilitate swallowing will also be used if and when needed. The children or their parents will be asked to fill in a food diary during one week after surgery.
  Interventions: Dietary Supplement: Timbal diet
- Extended telephone counseling (Other): Extended telephone counseling & Usual care : A nurse will contact the child, or the child´s parents, by telephone on day 1, 3, 5 and 10 for extended telephone counseling postoperatively (POD), to provide support and information. The child's well-being will be assessed, response given to queries and concerns, advice and explanations related to the problems expressed or identified, proper interventions will be promoted and reassurance provided. The nurse will fill in a protocol on what topics the counseling was about at each call and the child and/or parent a diary.
  Interventions: Other: Extended telephone counseling

INTERVENTIONS:
Combination Product: Acupuncture, acupressure — Intervention group will receive usual care in combination with Pyonex-needles and "Kulplåster". The control group will only receive usual care.
  Other Names: Pyonex-needles (Seirin, 1.5 mm long); "Kulplaster" (1.5 mm ball)
  Arms: Acupuncture, acupressure
Dietary Supplement: Timbal diet — Intervention group will receive usual care in combination Timbal diet including Protein-enriched ice cream, made with egg yolks and Cream. The control group will only receive usual care.
  Other Names: Protein-enriched ice cream, made with egg yolks and cream
  Arms: Timbal diet
Other: Extended telephone counseling — Intervention group will receive usual care in combination with Extended telephone counseling. The control group will only receive usual care.
  Arms: Extended telephone counseling

SUMMARY:
Children recovering from tonsil surgery following day surgery Tonsil surgery - self-care and treatment - the TONIST-study The main objective of this study is to evaluate the effect and experience of acupuncture, acupressure, specially designed diet and telephone counselling on children's surgery-related symptoms, quality of life and costs during recovery after tonsillectomy (TE) or tonsillotomy (TT).

Early discharge from hospitals means that patients have to deal with much of the post-operative care during recovery process on their own or with the help of relatives. The recovery period may be a progressive process of physical weakness (1,2).

In Sweden, 14 000 tonsil surgeries per year are performed, about 50% children under 15 years because of obstruction, of TE, tonsillectomy, and TT, tonsillomy. Children's tonsil surgery following day surgery are in focus for this study. Both qualitative and quantitative methods will be used.

DETAILED DESCRIPTION:
The TONIST-study

Acronyms:

APU Acupuncture, APR Acupressure, CReDECI Criteria for Reporting the Development and Evaluation of Complex Interventions in Healthcare, CG control group, IG intervention Group, PONV Postoperatively nausea and vomiting, PRiC Postoperative Recovery in Children, EQ5D EuroQol five dimensions' questionnaire

A pilot study will include evaluating the amount of issues in the instruments perceived possible to answer and/or the number of measurement points are reasonable.

Children's tonsil surgery following day surgery are in focus for this study. Children admitted for day surgery is monitored only a few hours after the surgery before going home when the parents must take the main responsibility for the care and monitoring during the recovery period (3). The present study design does not depend on the type of tonsil operation implemented, but the percentage advantage lodge will result in the description. Fifty percent of these surgical procedures are performed as day surgeries (4). The procedure causes a postoperative period of pain and risk of bleeding (5). The pain increases up to seven days after surgery, leading to problems with eating, drinking and sleeping (6). Children seem to receive too little analgesia and there seems to be a great need for postoperative information (7). Especially when the procedure is performed as day surgery the professional postoperative treatment at hospital is transferred to the patient to perform self-care. For the parents of young children, it could be a demanding task (8). Furthermore, the children's need of care could lead to loss of income since temporary parental benefit for care of the child will be necessary as well as absence from work and increased costs for the healthcare organization. Evidence-based interventions should constitute the basis for development of health care and post-operative interventions are often very complex, involving physical and emotional mechanisms. There is a gap in knowledge about effective interventions after tonsil surgery that could ease the self-care performed at home. In the proposed trials the investigators want to evaluate the effects of APU, APR, specially designed diet and extended telephone counselling on relieving common postoperative symptoms.

Qualitative and quantitative methods will be used. All the intervention groups will receive usual care in combination with a special intervention. The control group will receive usual care. The three interventions will be performed at one hospital each.

The investigators will apply "The new Medical Research Council Guidance" (9). Guidelines, CReDECI, will be used (10). In accordance with these criteria, reporting will be intersected in several publications; articles on the development, structured literature review and pilot testing, testing PRiC for children under 4 years and adolescents over 12 years, the evaluation of interventions and implementations.

Intervention I: Combinating APU and APR the investigators will evaluate the effect and safety as administered in clinical use which is a more holistic approach.

Intervention II: A specially designed diet including protein-enriched ice cream as snacks and "Timbalkost", specially designed diet, originally made for patients suffering of dysphagia will be used. "Timbalkost" will be given as lunch and dinner. Ice crème will be available as a snack, with lemon, vanilla and caramel flavor.

Intervention III: Extended telephone counseling. A nurse will contact the Child/youth, or the parents, by telephone on day 1, 3, 5 and 10 postoperatively, to provide support and information. The nurse will fill in a protocol on what topics the counseling was about at each call.

Usual care will be given to CG, and the IG. Usual care consists routines at the clinic, such as sedatives prior surgery, anesthesia during the operation and ondansetron and/or metoclopramide for PONV (11). For pain, paracetamol and NSAID is administered routinely postoperatively. Morphine is given intravenously in case of severe pain. Current standard care concerning diet is most often advice to eat and drink normally.

Participants Children, 2-19years of age who undergo TE or TT will be asked to participate.

Primary outcome is throat pain measured with the questionnaire PRiC, change is being assessed up to 21 days following surgery. The three interventions are to be evaluated with registration of postoperatively recovery.

The primary outcome will be measured by PRiC regarding existing pain in the throat (12). Regarding pain, the child could in the enquiry choose one of four options; During the last day/night (within the last 24 hours) Have I had a sore throat with the opportunity to grade the answer Not at all, A little, alternatively Much or Very much.

Estimates for the number of children who need to be included in the study is based on the distribution of responses to the question "sore throat" that is, a sore throat the last 24 hours from the questionnaire PRiC. The control group is assumed to respond to the same distribution as the children in Bramhagen et al (12) and the children in the intervention group is assumed to have a positive shift in the distribution of answers as shown below, where 1 = Not at all throat pain, 2 = Little hurt throat, 3=Very sore throat or 4 = Very much sore throat.

A positive shift in response to previous study results in Bramhagen (12) is assumed in the Intervention Group.

In order to statistically ensure a difference between the intervention and control based on the conditions above, you need 138 children in each of the four groups, a total of 828 children. The method used is the Mann Whitney U test with 80% power and 5% alpha.

Secondary outcomes; change is being assessed following the surgery. The secondary outcome is any change in nausea, vomiting and other parts of the questionnaire PRiC. Analyzes regarding costs will be carried out both in a social and a medical perspective. Outcome after different types of surgery may emerge. The economic effects will be evaluated between IG and CG and between the interventions. Children and parent's experiences after surgery will be monitored through qualitative interviews. An economic evaluation of the three interventions combined with parents' absence from work will be made (IG and CG). Quality of life, including health-related status will be measured using EQ5D (questionnaire for health) (13).

Data collection for registration of the children' recovery from their surgery the instruments Postoperative Recovery in Children instrument (PRiC) (12) will be used in each Cg and IG.

PRiC is based on data about the general recovery of postoperative symptoms such as pain in the throat, including information on the various physical and emotional symptoms. PRiC is measured on a four-point scale children's signs and symptoms during the last day/night in the last 24 hours, not at all, a little, a lot or very much. It is questioned, for example, "I felt as if I would vomit, I have had vomiting, I have had a sore throat or had blood in my mouth." It is also requested for the child "I have found it difficult to eat, I have found it difficult to play/be active or have I found it difficult to attend daycare/school. Finally, the questionnaire asks about" Right now I feel very good, fairly good, quite bad or very bad (12).

For measuring pain, nausea and anxiety at baseline i.e. before surgery, preoperately the Numerical rating scale (NRS) will be used, asking the nurse to document in the child's medical record. The Investigators will seek to gain access to the child's medical record. The instruments will be used collecting data according to the time schedule (Table 2) in both IG and CG and with help from the parents if needed. PRiC will be used on the day of surgery and thereafter assessed over time following the surgery daily on postoperative days 1-7 the postoperative days 10, 14, 21. EQ5D will be measures at baseline 14 Days Before surgery and thereafter assessed over time on postoperative days 10, 14 and 21. Diary for Specially designed diet will be assessed over time daily following surgery as long as the Child use the diet. Protocol and diary for telephone follow up will be assessed over time following surgery on postoperative days 1, 3, 5 and 10. Diary for APU and APR will be assessed over time following surgery on the surgery day and daily the postoperative days 1-10.

Measuring time points:

Numerical rating scale NRS (0-10) pain, nausea and anxiety measured before premedication on surgery day.

PRiC, recovery measured on surgery day, daily following surgery on days 1-7 and on days 10, 14, 21 following surgery.

EQ5D, Quality of life and health measured 14 days before surgery, postoperative days 10, 14 and 21 following surgery.

Diary for Specially designed diet Experience and number of meals measured up to 7 days after surgery.

Protocol and diary for telephone follow up. Documentation of given support and on the postoperative days 1, 3, 5 and up to day 10 postoperatively.

Protocol and diary for APU and APR Documentation of when APU and APR were used for any reason and when removed. Documentation daily on surgery day and postoperative days 1-10.

The diaries on needle stimulation and the food will be collected after one week, data on the telephone calls after 10 days in the IG:s. For each patient specific operation data will be collected on day one and postoperative complications after 30 days and 6 months, in the child´s medical records and in the Swedish Tonsil register.

The economic evaluations: EQ5D, data about patients' contacts with healthcare professionals and the parents' number of days they are absent from work. Data on indication for surgery, surgical techniques and hemostasis method will be collected from the children's medical record at baseline and any postoperative complications within 6 months.

Ten children (or parents if the child is younger than 15 years of age) in each IG and the CG will be interviewed using open questions at POD 14 (60 interviews in total) about their experiences of the respectively IG or CG.

The quantitative data will be analyzed using relevant statistical methods (Altman 2006). Depending on type of data and distribution either parametric (ANOVA) or non-parametric assays to assess group differences. For analysis of binary outcome measures the investigators will apply logistic regression models.

The interviews will be transcribed and analyzed using content analysis (14) with an inductive approach to illuminate children's/parents' experiences.

ELIGIBILITY:
Inclusion Criteria: Children, 2-19 years of age who undergo Tonsillectomy or Tonsillotomi be asked to participate.

Exclusion Criteria:

For children who have aversion, intolerance or allergy to ice cream or any of the ingredients in it the exclusion of the ice cream as a snack will be done.

Ages: 2 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 576 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Sore throat item, in the instrument Postoperative Recovery in Children instrument (PRiC), change assessed | On the surgery day, Daily during the postoperative days 1-7 and during the 10:th, 14:th and the 21:th day
  Sore throat measured with the PRiC, instrument. Sore throat with the opportunity to grade the answer Not at all, A little, alternatively Much or Very much.
  Estimates for the number of children who need to be included in the study is based on the distribution of responses to the question "sore throat" that is, a sore throat the last 24 hours from the questionnaire PRiC. The control group is assumed to respond to the same distribution as the children in Bramhagen et al (2016) and the children in the intervention group is assumed to have a positive shift in the distribution of answers.

SECONDARY OUTCOMES:
Numerical Rating Scale, NRS (0-10) Nausea | Baseline, before premedication before the surgey starts i.e. preoperative and on postopertive day 2
  Nausea on a scale NRS (0-10)
Postoperative Recovery in Children, PRiC, Questionaire. | Daily during the postoperative days 1-7 and during the 10:th, 14:th and the 21:th day
  Measuring change in postoperative recovery in children emotional state.
EQ5D Economic effect between, assessment of change | On the 14:th day before surgery, Daily during the 10:th, 14:th and the 21:th postoperative days
  Quality of life and health
Protocol and diary for telephone follow up, assessment of change | On the first postoperative day and on the 3:rd, 5:th och 10:th day postoperatively.
  postoperative problems that arise, assessment of these and reference to the healthcare institution if necessary
Diary for acupuncture and acupressure, assessment of change | On the surgery day and daily on the postoperative days 1 to at 10. Measurement to the high tenth day postoperatively depending on whether the child is using the APU and / or LFS for so long.
  Documentation of when akupunkture or acupressure is given , for what reason and when removed
Diary for specially designed diet including ice Cream, assessment of change | As long as meals are consumed, daily, up to 10 days following surgery day.
  Diary documentation, number of meals.
Numerical Rating Scale, NRS (0-10) anxiety | Baseline, before premedication before the surgey starts i.e. preoperative and on postopertive day 2
  Anxiety on a scale NRS (0-10)
Numerical Rating Scale, NRS (0-10) | Baseline, before premedication before the surgey starts i.e. preoperative and on postopertive day 2
  Pain on a scale NRS (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Helena i Rosén, PhD, Principal Investigator — Health scienses, Faculty of medicine, Lund University; Lena-karin Erlandsson, PhD, Study Director — Health scienses, Faculty of medicine, Lund University
Locations (1):
- Helena Rosén, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allvin R, Berg K, Idvall E, Nilsson U. Postoperative recovery: a concept analysis. J Adv Nurs. 2007 Mar;57(5):552-8. doi: 10.1111/j.1365-2648.2006.04156.x. PMID 17284272
- [Background] Jakobsson, J. (2017). The process of recovery after colorectal cancer surgery : patients' experiences and factors of influence. Malmö högskola. Fakulteten för hälsa och samhälle, Malmö University Doctoral Dissertation: 93.
- [Background] Young, J., et al. (2000). Day surgery patients' convalescence at home: Does enhanced discharge education make a difference? Nursing & Health Sciences 2(1): 29-39.
- [Background] Stalfors, J. (2015). Registerdata från Öron-, Näs- och Hals kvalitetsregister (2015) PDF Rapport ISSN 1400-0121 SVENSK ÖNH-TIDSKRIFT 22(3).
- [Background] Ericsson, Elisabeth. (2007). Health and well-being of children and young adults in relation to surgery of the tonsils. (Medical dissertation), Linköping University Linköping, Sweden. (No. 992.)
- [Background] Stanko D, Bergesio R, Davies K, Hegarty M, von Ungern-Sternberg BS. Postoperative pain, nausea and vomiting following adeno-tonsillectomy - a long-term follow-up. Paediatr Anaesth. 2013 Aug;23(8):690-6. doi: 10.1111/pan.12170. Epub 2013 May 13. PMID 23668258
- [Background] Paquette J, Le May S, Lachance Fiola J, Villeneuve E, Lapointe A, Bourgault P. A randomized clinical trial of a nurse telephone follow-up on paediatric tonsillectomy pain management and complications. J Adv Nurs. 2013 Sep;69(9):2054-65. doi: 10.1111/jan.12072. Epub 2013 Jan 13. PMID 23311981
- [Background] Sutters KA, Savedra MC, Miaskowski C. The pediatric PRO-SELF(c): pain control program: an effective educational program for parents caring for children at home following tonsillectomy. J Spec Pediatr Nurs. 2011 Oct;16(4):280-94. doi: 10.1111/j.1744-6155.2011.00299.x. Epub 2011 Aug 12. PMID 21951354
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Background] Mohler R, Kopke S, Meyer G. Criteria for Reporting the Development and Evaluation of Complex Interventions in healthcare: revised guideline (CReDECI 2). Trials. 2015 May 3;16:204. doi: 10.1186/s13063-015-0709-y. PMID 25935741
- [Background] Segerdahl M, Warren-Stomberg M, Rawal N, Brattwall M, Jakobsson J. Children in day surgery: clinical practice and routines. The results from a nation-wide survey. Acta Anaesthesiol Scand. 2008 Jul;52(6):821-8. doi: 10.1111/j.1399-6576.2008.01669.x. Epub 2008 May 21. PMID 18498436
- [Background] Bramhagen AC, Eriksson M, Ericsson E, Nilsson U, Harden S, Idvall E. Self-reported post-operative recovery in children: development of an instrument. J Eval Clin Pract. 2016 Apr;22(2):180-8. doi: 10.1111/jep.12451. Epub 2015 Oct 13. PMID 26460499
- [Background] Dolan P. Modeling valuations for EuroQol health states. Med Care. 1997 Nov;35(11):1095-108. doi: 10.1097/00005650-199711000-00002. PMID 9366889
- [Background] Graneheim UH, Lundman B. Qualitative content analysis in nursing research: concepts, procedures and measures to achieve trustworthiness. Nurse Educ Today. 2004 Feb;24(2):105-12. doi: 10.1016/j.nedt.2003.10.001. PMID 14769454
- [Derived] Gudnadottir G, Persson RG, Drevenhorn E, Olofsson E, Rosen H. The effect of telephone counseling and internet-based support on pain and recovery after tonsil surgery in children - a systematic review. Int J Nurs Stud Adv. 2021 Apr 22;3:100027. doi: 10.1016/j.ijnsa.2021.100027. eCollection 2021 Nov. PMID 38746736